CLINICAL TRIAL: NCT06007573
Title: Acupuncture Combined With Nimodipine for Prevention of Post-stroke Dementia:a Randomized Controlled Trial
Brief Title: Acupuncture Combined With Nimodipine for Prevention of Post-stroke Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzhen Pan (Other)
Collaborators: Department of acupuncture and massage, Nanling Hospital of traditional Chinese Medicine, Nanling County, Wuhu City, Anhui Province (Unknown)
Responsible Party: Sponsor-Investigator, Yuzhen Pan, DOCTOR, The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Organization: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-zj-21
Record Dates: First submitted 2023-08-15; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Post-stroke Dementia
Keywords: randomized controlled trial; post-stroke dementia; Acupuncture; nimodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): On the basis of the control group treatment, the treatment group also adopted the acupuncture treatment
  Interventions: Drug: The control group received oral nimodipine tablets
- control group (Other): The control group received oral nimodipine tablets
  Interventions: Drug: The control group received oral nimodipine tablets

INTERVENTIONS:
Drug: The control group received oral nimodipine tablets — The control group received oral nimodipine tablets

SUMMARY:
To observe the clinical efficacy of TCM acupuncture combined with western medicine nimodipine for prevention of post-stroke dementia by comparing with clinical conventional treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. Definite ischemic stroke or hemorrhagic stroke confirmed by head CT / MRI examination
2. Memory or cognitive and executive dysfunction. Cognitive dysfunction will be determined after the mini mental state evaluation (MMSE) score
3. Age limited to 40-85 years, irrespective of gender
4. Stable condition, clear consciousness, no aphasia, oral medication available
5. No major comorbidity, no major depression
6. Consent and signed patient informed consent

Exclusion Criteria:

1. Had serious medical conditions, such as heart, liver, kidney, or endocrine disease
2. Aphasia or hearing impairment
3. Participants in other clinical trials
4. Patients currently on medication to improve cognitive function

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Response Rate | 24 weeks

SECONDARY OUTCOMES:
Hasegawa Dementia Scale | 24 weeks
Montreal Cognitive Assessment | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui University of Chinese Medicine, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
At present, we have not made a decision on whether to share all IPD. This is because we need to consider a range of factors, including ethical principles, legal requirements, privacy protection, and data sharing agreements. We are carefully evaluating these factors and will make a clear decision as soon as possible.